CLINICAL TRIAL: NCT06689800
Title: Let's Get REAL: A Pilot Trial of a Family Health Communication Tool in Pediatric Stem Cell Transplant and Cellular Therapy
Brief Title: Let's Get REAL: Family Health Communication Tool in Pediatric Stem Cell Transplant and Cellular Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202410119; K12CA167540 (NIH)
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Malignancy; Solid Tumor; Sickle Cell Disease; Aplastic Anemia; Immune Deficiency; Metabolic Disorder
Keywords: Pediatric; Family; Decision making; Health Communication; Intervention
MeSH Terms: conditions — Hematologic Neoplasms; Anemia, Sickle Cell; Anemia, Aplastic; Immunologic Deficiency Syndromes; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Let's Get REAL family health communication tool: Patients (8-12 years of age) (Experimental): Patients and parent(s) will be given the Let's Get REAL family health communication tool to use up to one month prior to their SCTCT consultation visit. It is a guide for pediatric patients and their families to learn about and discuss SCTCT. Participants will complete demographic and baseline surveys prior to using the tool, and then additional surveys up to one month after SCTCT consultation visit and up to one month post-discharge from SCTCT. SCTCT consultation visits will be audio-recorded. Participants may also participate in an optional semi-structured interview up to 8 weeks after SCTCT consultation.
  Interventions: Behavioral: Let's Get REAL
- Let's Get REAL family health communication tool: Patients (13-17 years of age) (Experimental): Patients and parent(s) will be given the Let's Get REAL family health communication tool to use up to one month prior to their SCTCT consultation visit. It is a guide for pediatric patients and their families to learn about and discuss SCTCT. Participants will complete demographic and baseline surveys prior to using the tool, and then additional surveys up to one month after SCTCT consultation visit and up to one month post-discharge from SCTCT. SCTCT consultation visits will be audio-recorded. Participants may also participate in an optional semi-structured interview up to 8 weeks after SCTCT consultation.
  Interventions: Behavioral: Let's Get REAL
- Let's Get REAL family health communication tool: Parents (Experimental): Patients and parent(s) will be given the Let's Get REAL family health communication tool to use up to one month prior to their SCTCT consultation visit. It is a guide for pediatric patients and their families to learn about and discuss SCTCT. Participants will complete demographic and baseline surveys prior to using the tool, and then additional surveys up to one month after SCTCT consultation visit and up to one month post-discharge from SCTCT. SCTCT consultation visits will be audio-recorded. Participants may also participate in an optional semi-structured interview up to 8 weeks after SCTCT consultation.
  Interventions: Behavioral: Let's Get REAL

INTERVENTIONS:
Behavioral: Let's Get REAL — Family health communication tool

SUMMARY:
The investigators will conduct a pilot feasibility and efficacy trial of a newly developed family health communication tool (called Let's Get REAL) in increasing youth involvement in real-time stem cell transplant and cellular therapy decisions (SCTCT). The investigators will pilot the intervention among 24 youth and their parents, stratified by youth age (stratum 1, 8-12 years of age and stratum 2, 13-17 years of age).

ELIGIBILITY:
Inclusion Criteria Youth:

* Children or adolescents 8-17 years of age referred for SCTCT.
* Diagnosis of malignant or nonmalignant disorder.
* Referred for any type of SCTCT. Autologous and allogeneic stem cell and cellular therapies are eligible.
* Planning to meet with a provider to discuss SCTCT.
* Must have the ability to understand and willingness to consent to participate after reviewing an IRB approved informed assent document.
* Must speak English and be cognitively able to participate.

Inclusion Criteria Parents:

* Parent or guardian of a child 8-17 years of age with any diagnosis referred for any type of SCTCT. Diagnoses may include malignant and nonmalignant disorders. Autologous and allogeneic stem cell and cellular therapies are eligible. Parent or guardian is defined as an adult who usually cares for the youth and has authority to make medical decisions for them.
* Must have the ability to understand and willingness to consent to participate after reviewing an IRB approved informed consent document.
* Must speak English and be cognitively able to participate.

Exclusion Criteria Youth:

* Active medical problems severe enough to preclude study participation at the time of recruitment.

  * Patients who are otherwise eligible, but whose primary transplant physician does not want them to participate in the study.
* Lacks cognitive capacity to complete study activities, as determined by consenting professional.

Exclusion Criteria Parents:

* Their youth referred for SCTCT does not assent to participate.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intervention as measured by the Feasibility of Intervention questionnaire | Up to 4 weeks after SCTCT consultation (estimated to be week 8)
  This is a 4-item scale that youth and their parents report feasibility of the intervention on a 5-point Likert scale ranging from 'Completely disagree' to Completely agree'. A higher score indicates greater feasibility.
Acceptability of intervention as measured by the Acceptability of Intervention questionnaire | Up to 4 weeks after SCTCT consultation (estimated to be week 8)
  This is a 4-item scale that youth and their parents report acceptability of the intervention on a 5-point Likert scale ranging from 'Completely disagree' to Completely agree'. A higher score indicates greater acceptability.
Appropriateness of intervention as measured by the Intervention of Appropriateness questionnaire | Up to 4 weeks after SCTCT consultation (estimated to be week 8)
  This is a 4-item scale that youth and their parents report appropriateness of the intervention on a 5-point Likert scale ranging from 'Completely disagree' to Completely agree'. A higher score indicates greater appropriateness.
Feasibility of intervention as measured qualitatively | Up to 8 weeks after SCTCT consultation (estimated to be week 16)
  Content analysis of open-ended survey responses and quotations from individual interviews. Will be collecting number of feasibility content codes.
Acceptability of intervention as measured qualitatively | Up to 8 weeks after SCTCT consultation (estimated to be week 16)
  Content analysis of open-ended survey responses and quotations from individual interviews. Will be collecting number of acceptability content codes.
Appropriateness of intervention as measured qualitatively | Up to 8 weeks after SCTCT consultation (estimated to be week 16)
  Content analysis of open-ended survey responses and quotations from individual interviews. Will be collecting number of appropriateness content codes.

SECONDARY OUTCOMES:
Difference in feasibility scores in those 8-12 years of age and those 13-17 years of age as measured by the Feasibility of Intervention questionnaire | Up to 4 weeks after SCTCT consultation (estimated to be week 8)
  This is a 4-item scale that youth and their parents report feasibility of the intervention on a 5-point Likert scale ranging from 'Completely disagree' to Completely agree'. A higher score indicates greater feasibility.
Difference in acceptability scores in those 8-12 years of age and those 13-17 years of age as measured by the Acceptability of Intervention questionnaire | Up to 4 weeks after SCTCT consultation (estimated to be week 8)
  This is a 4-item scale that youth and their parents report acceptability of the intervention on a 5-point Likert scale ranging from 'Completely disagree' to Completely agree'. A higher score indicates greater acceptability.
Difference in appropriateness scores in those 8-12 years of age and those 13-17 years of age as measured by the Intervention of Appropriateness questionnaire | Up to 4 weeks after SCTCT consultation (estimated to be week 8)
  This is a 4-item scale that youth and their parents report appropriateness of the intervention on a 5-point Likert scale ranging from 'Completely disagree' to Completely agree'. A higher score indicates greater appropriateness.
Perceived levels of decision-making involvement in youth 8-17 years of age and their parents as measured by the Decision Making Involvement Scale | Up to 4 weeks after SCTCT consultation (estimated to be week 8)
  This is a 30-item scale that youth and their parents report youth involvement behaviors in a decision related to their illness on a 4-point Likert scale ranging from 'A Little Bit' to 'A Lot'. The higher the subscale score (child seek, child express, parent seek, parent express, and joint/options), the more that behavior or type of involvement occurred in the decision making process.
Observed levels of decision-making involvement in youth 8-17 years of age and their parents | Up to 4 weeks after SCTCT consultation (estimated to be week 8)
  Number of utterance occurrences for the following: 1) who uttered (youth, parent), 2) was utterance prompted (yes/no), if so, by who, 3) type of utterance (questions, opinion, concern, other), and 4) content of utterance (prognosis, side effect, expectation).
Change in youth-parent communication as measured by the Likert-type Parent-Adolescent Communication Scale | Up to 4 weeks prior to SCTCT consultation and up to 4 weeks after SCTCT consultation (estimated to be 8 weeks)
  This is a 20-item scale that youth and parents report the degree of openness in family communication and the extent of problems with family communications on a 5-point Likert ranging from 'strongly disagree' to 'strongly agree'. A higher score on the degree of openness subscale indicates better communication between parent and adolescent. For extent of problems subscale, a higher score indicates more problems in the parent-child communication.
Change in the level of youth's general anxiety as measured by the Likert-type PROMIS Anxiety 8a Short Form or parent proxy | Up to 4 weeks prior to SCTCT consultation and up to 4 weeks after SCTCT consultation (estimated to be 8 weeks)
  This is an 8-item scale that measures youth's general anxiety in those 8-17 years of age on a 5-point Likert scale ranging from 'never' to 'almost always'.
Level of decisional conflict as measured by the Likert-type Decisional Conflict Scale | Up to 4 weeks after SCTCT consultation (estimated to be week 8)
  This is a 10-item scale that youth and parents report their personal uncertainty and decisional conflict related to a specific decision. We are using the question format as it is recommended for those with limited reading or response skills. They respond 'Yes', 'No, or 'Unsure'. A total decision conflict score ranges from 0 (no decisional conflict) to 100 (extremely high decision conflict). Higher scores on subscales uncertainty, informed, values clarity, and support reflect feeling extremely uncertain about the best choice, feeling extremely uninformed, feeling extremely unclear about personal values, and feeling extremely unsupported in decision making respectively.
Youth-parent congruence of youth decision making involvement as measured by two Likert type statements | Up to 4 weeks after SCTCT consultation (estimated to be week 8)
  Number of dyads that agree on these two statements measured on a 4-point Likert scale ranging from 'Not at all' to 'A lot': 1)"I/my child should be involved in future talks about transplant" and 2) "I/my child wants to be involved in future talks about transplant".
Satisfaction with the decision making involvement as measured by one Likert type statement | Up to 4 weeks after SCTCT consultation (estimated to be week 8)
  This is a one item statement, "I am satisfied with my/my child's involvement in the transplant decision making process", measured on a 4-point Likert scale ranging from 'Not at all' to 'A lot'. A higher score indicates more satisfaction.
Number of patients who chose SCTCT | Up to 4 weeks after SCTCT consultation (estimated to be week 8)

CONTACTS AND LOCATIONS:
Overall Officials: Ginny Schulz, Ph.D., RN, CPNP-PC, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu